CLINICAL TRIAL: NCT02863445
Title: Improving the Effectiveness of Orally Dosed Emergency Contraceptives in Obese Women - Pharmacodynamics of 3.0mg LNG
Brief Title: Effectiveness of Orally Dosed Emergency Contraception in Obese Women - LNG
Acronym: EC-Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Alison Edelman, Professor, OB/GYN, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB 16291
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Obesity; Body weight; Emergency contraception; Levonogestrel; Ulipristal acetate
MeSH Terms: conditions — Obesity; Body Weight | interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LNG-ECx1 (Active Comparator): Levonorgestrel 1.5 mg orally x 1 dose. Timing of dosage depends on ovarian follicle measurements.
  Interventions: Drug: Levonorgestrel-based emergency contraception 1.5 mg
- LNG-ECx2 (Experimental): Levonorgestrel 3mg orally x 1 dose. Timing of dosage depends on ovarian follicle measurements.
  Interventions: Drug: Levonorgestrel-based emergency contraception 3.0mg

INTERVENTIONS:
Drug: Levonorgestrel-based emergency contraception 1.5 mg — Evaluating pharmacodynamic outcomes in obese women using 1.5mg versus 3.0mg of LNG-based EC
  Other Names: Plan B; Next Choice
  Arms: LNG-ECx1
Drug: Levonorgestrel-based emergency contraception 3.0mg — Evaluating pharmacodynamic outcomes in obese women using 1.5mg versus 3.0mg of LNG-based EC
  Arms: LNG-ECx2

SUMMARY:
Obese women are significantly more likely than their normal BMI counterparts to experience failure of orally-dosed emergency contraceptives. The PI's preliminary data provides evidence for testing a dose escalation strategy in an effort to provide improved efficacy from orally-dosed emergency contraceptives in obese women. The overall project will be focused on both levonorgestrel (LNG) - and ulipristal acetate-containing emergency contraception but this protocol registration is for the LNG aspect of the study procedures.

DETAILED DESCRIPTION:
Emergency contraception (EC) provides a woman with an additional line of defense against unintended pregnancy following an act of unprotected intercourse. Orally-dosed EC works by delaying ovulation and reduces the risk of pregnancy for a single act of unprotected intercourse by 50-70%. Unfortunately, obese women are significantly more likely than their normal BMI counterparts to experience failure of orally-dosed EC and in some instances EC is equivalent to placebo.

The PI's preliminary data provides evidence for testing a dose escalation strategy in an effort to provide improved efficacy from orally-dosed EC in obese women. The hypothesis is that increasing the dose of orally-dosed EC agents will normalize the pharmacokinetics resulting in the expected treatment effect (delay in follicle rupture) in obese women. In the overall proposal, the investigators plan to perform detailed pharmacokinetic and pharmacodynamic studies of ulipristal acetate-based EC in obese women and expand upon the preliminary findings of levonorgestrel-based EC. This protocol registration is for the LNG aspect of the study procedures focused on the pharmacodynamics of LNG dose escalation

ELIGIBILITY:
Inclusion Criteria:

* Generally health women
* Aged 18-35 years old
* Regular menses (every 21-35 days) experiencing an ovulatory screening cycle with a progesterone level of 3ng/ml or greater.
* Subjects must have a BMI of >30 kg/m2 and weigh at least 80 kg or more.

Exclusion Criteria:

* Metabolic disorders including uncontrolled thyroid dysfunction and Polycystic Ovarian Syndrome
* Impaired liver or renal function
* Actively seeking or involved in a weight loss program (must be weight stable) pregnancy, breastfeeding, or seeking pregnancy
* Recent (within last 8 weeks) use of hormonal contraception
* Current use of drugs that interfere with metabolism of sex steroids
* Smokers.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
PI acknowledges willingness to share data and materials with other investigators through established means. Data will be shared with collaborators as soon as available; with other scientists before publication if the work to be done is different from the PI's purposes; with local colleagues at seminars and talks including the yearly university-wide research-in-progress seminar; and with the scientific community at large by posters and presentations at local, regional, national, and international scientific meetings. Data will be presented via publication to the widest audience possible.
  Transfer of resources is subject to the acceptance of a Materials Transfer Agreement as required by policy at OHSU.
  OHSU complies with NIH policy on Sharing Research Data and on Sharing Model Organisms.

REFERENCES:
- [Background] Edelman AB, Cherala G, Blue SW, Erikson DW, Jensen JT. Impact of obesity on the pharmacokinetics of levonorgestrel-based emergency contraception: single and double dosing. Contraception. 2016 Jul;94(1):52-7. doi: 10.1016/j.contraception.2016.03.006. Epub 2016 Mar 18. PMID 27000996
- [Result] Edelman AB, Hennebold JD, Bond K, Lim JY, Cherala G, Archer DF, Jensen JT. Double Dosing Levonorgestrel-Based Emergency Contraception for Individuals With Obesity: A Randomized Controlled Trial. Obstet Gynecol. 2022 Jul 1;140(1):48-54. doi: 10.1097/AOG.0000000000004717. Epub 2022 Jun 7. PMID 35849455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at Oregon Health & Science University and Eastern Virginia Medical School from June 2017 to February 2021. The study recruited healthy individuals aged 18-35 years with regular menstrual cycles (21-35 days) and BMIs higher than 30 with weights of 176 pounds or more.
Pre-assignment Details: After enrollment, participants started their treatment cycle at the time of next menses or could delay for 1-2 menstrual cycles if a scheduling conflict occurred. On days 6-8 of the treatment cycle, participants were monitored every other day for follicular activity with transvaginal ultrasonographic examination, as well as blood sampling for progesterone, estradiol, and LH until a dominant follicle measuring 15 mm or greater in at least one dimension was visualized.
Period: Overall Study
Arm/Group | LNG-ECx1 | LNG-ECx2
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants completed the study and were part of the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | LNG-ECx1 | LNG-ECx2 | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (3.5) | 29.3 (4.4) | 28.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 28 | 30 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 27 | 27 | 54
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Nulligravid [Count of Participants; unit: Participants] | 16 | 19 | 35
BMI [Mean (Standard Deviation); unit: kg/m^2] | 37.3 (5.4) | 38.8 (5.8) | 38.0 (5.6)
Weight (lbs) [Mean (Standard Deviation); unit: pounds] | 224.9 (33.1) | 236.4 (39.1) | 230.7 (36.5)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants in Two Treatment Groups (1.5mg Levonorgestrel and 3mg Levonorgestrel) With no Follicle Rupture at 5 Days Within One Menstrual (Treatment) Cycle.
Description: No evidence of follicle rupture achieved by participant in one menstrual (treatment) cycle at 5 days post LNG dosing. Follicle rupture is defined as the disappearance of or >50% reduction in the size of the leading follicle. Dosing occurred after a dominant follicle measuring 15 mm or greater in at least one dimension was visualized on ultrasound.
Time Frame: 5 days post-LNG dosing
Measure: Number; unit: participants
Arm/Group | LNG-ECx1 | LNG-ECx2
Number analyzed (Participants) | 35 | 35
participants | 18 | 24

2. Secondary Outcome: Number of Participants With Follicle Rupture Before 5 Days
Description: Among the participants with follicle rupture before 5 days, the time to rupture was measured and reported for each day up to day 5. If the date of follicle rupture was unclear by ultrasonographic imaging (eg, collapse was seen, but reduction of size was less than 50%), serum hormone levels were used to adjudicate day of ruptures.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | LNG-ECx1 | LNG-ECx2
Number analyzed (Participants) | 35 | 35
Participants | 17 | 11

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | LNG-ECx1 | LNG-ECx2
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 13/35 | 14/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNG-ECx1 (N=35) | LNG-ECx2 (N=35)
Menstrual Cramping (Reproductive system and breast disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 3 | 6
Headache (Nervous system disorders) | 1 | 2
Common Cold (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Abdominal Cramping (General disorders) | 2 | 2
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT02863445/Prot_SAP_000.pdf